CLINICAL TRIAL: NCT00232531
Title: Cardiovascular Magnetic Resonance Evaluation of the Effects of Niaspan on Regression of Atherosclerosis and Restoration of Endothelial Function
Brief Title: Oxford Niaspan Study: Effects of Niaspan on Atherosclerosis and Endothelial Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Oxford (Other)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 04.OXA.020
Record Dates: First submitted 2005-10-03; First posted 2005-10-04 (Estimated); Last update posted 2007-01-29 (Estimated); Status verified 2006-09

CONDITIONS: Atherosclerosis
MeSH Terms: conditions — Atherosclerosis | interventions — Niacin

INTERVENTIONS:
Drug: Niaspan

SUMMARY:
AIM 1 will test the hypothesis that elevation of high-density lipoprotein (HDL) through treatment with Niaspan will accelerate the regression of atherosclerotic plaque in patients with established atherosclerosis. The investigators will therefore study patients with atherosclerosis in the aorta and carotid artery. Plaque quantification will be with magnetic resonance imaging (MRI).

AIM 2 will assess the ability of Niaspan to improve endothelial function in patients with coronary artery disease and type II diabetes mellitus, who typically have low high-density lipoprotein cholesterol (HDL-C), and high risk of cardiovascular events.

DETAILED DESCRIPTION:
Patients will be randomised to receive either Niaspan 2000mg each night or placebo. Niaspan will be commenced at 375mg daily and increased to 500mg then to 750, and 1000mg daily at weekly intervals. After 4 weeks the dose will be increased to 1500mg daily and, after a further one month, the study dose of 2000mg daily2 will be instigated. Immediately before randomization (to exclude patients unable to tolerate MRI because of claustrophobia), and 6 and 12 months after commencing treatment participants will undergo MR examination.

ELIGIBILITY:
Inclusion Criteria:

* Aim 1: Carotid or peripheral arterial disease and HDL <1mmol/L
* Aim 2: Coronary artery disease, type II diabetes and HDL <1mmol/L

Exclusion Criteria:

The following will constitute exclusion criteria:

* Inability to provide informed consent,
* Known intolerance of a study drug,
* Use of niacin or a fibrate at time of screening,
* AST or ALT elevated above normal range at time of screening
* Use of oral nitrates or nicorandil
* Uncontrolled or newly diagnosed diabetes mellitus
* Symptomatic heart failure or heart failure requiring treatment with diuretics
* Fasting triglycerides > 500mg/dL [5.65mmol/L]
* Patients with acute coronary syndromes, active peptic ulcer disease,
* Active gout,
* Standard exclusions for MRI will apply, i.e. pacemakers, implantable defibrillators, metal implants or embedded metallic fragments of any kind.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70
Dates: Start 2004-09; Study Completion 2009-02

PRIMARY OUTCOMES:
Regression of artheriosclerotic plaque measured using functional magnetic resonance imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Robin P Choudhury, DM, MRCP, Principal Investigator — University of Oxford
Locations (1):
- Oxford University, Oxford, United Kingdom

REFERENCES:
- [Derived] Lee JM, Robson MD, Yu LM, Shirodaria CC, Cunnington C, Kylintireas I, Digby JE, Bannister T, Handa A, Wiesmann F, Durrington PN, Channon KM, Neubauer S, Choudhury RP. Effects of high-dose modified-release nicotinic acid on atherosclerosis and vascular function: a randomized, placebo-controlled, magnetic resonance imaging study. J Am Coll Cardiol. 2009 Nov 3;54(19):1787-94. doi: 10.1016/j.jacc.2009.06.036. PMID 19874992